CLINICAL TRIAL: NCT00689598
Title: Use of Spironolactone to Treat Patients With Paroxysmal Atrial Fibrillation- A Multi-Center, Prospective, Randomized, Placebo-Controlled, Double Blind Study
Brief Title: Spironolactone for Paroxysmal Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Tsu-Juey Wu, M.D./Staff Physician, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C07061
Record Dates: First submitted 2008-03-30; First posted 2008-06-03 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation, spironolactone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- III (Placebo Comparator): Placebo
  Interventions: Drug: Spironolactone
- Experimental (Experimental): Drug intervention
  Interventions: Drug: Spironolactone; Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 25 mg po qd 25 mg po bid
  Other Names: Aldactone
Drug: Placebo — Spironolactone 25 mg po qd
  Other Names: Aldactone
  Arms: Experimental

SUMMARY:
To determine whether or not spironolactone can prevent or delay the occurrence of atrial fibrillation.

DETAILED DESCRIPTION:
To determine whether or not adding spironolactone can prevent or delay the occurrence of paroxysmal atrial fibrillation in patients who have received propafenone treatment.

ELIGIBILITY:
Inclusion criteria:

1. 18 to 80 Y/O,
2. Paroxysmal AF.

Exclusion criteria:

1. GPT>100 IU/L or tota bilirubin >2 mg/dl;
2. Creatinine > 2 mg/dl;
3. Serum potassium >= 5 mM;
4. Serum sodium <=130 mM;
5. Uric acid > 10 mg/dl。

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
time to a first electrocardiographically confirmed AF | 3 months

SECONDARY OUTCOMES:
1. Response rate: Improvement of any symptom scores and/or SF36 scores more than 50 % (compared with re-randomization scores) 2. Difference of mean episodes of documented AF between the spironolactone and placebo groups. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tsu-Juey Wu, M.D., Principal Investigator — TCVGH
Locations (1):
- Taichung General Hospital, Taichung, Taiwan